CLINICAL TRIAL: NCT03206723
Title: Bandage Contact Lenses to Decrease Pain and Improve Healing in Emergency Department Subjects Presenting With Corneal Abrasions
Brief Title: Bandage Contact Lenses for Corneal Abrasions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, David Tanen, Professor of Clinical X, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30610-01
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Corneal Abrasion; Eye Trauma
Keywords: corneal abrasion; contact lens; eye trauma
MeSH Terms: conditions — Corneal Injuries; Eye Injuries | interventions — Ophthalmic Solutions; Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Active Comparator): 1. Standard care
  Interventions: Drug: Eyedrop; Drug: Hydrocodone
- Group 2 (Active Comparator): 1. Standard care
  2. Bandage contact lens
  Interventions: Device: Bandage contact lens; Drug: Eyedrop; Drug: Hydrocodone

INTERVENTIONS:
Device: Bandage contact lens — Bandage contact lenses (BCL) have the advantage of pain reduction, facilitating epithelial healing, and improved surface healing. They have been used in the ophthalmology community to treat post-operative eye pain due to the large corneal abrasion created during Excimer photorefractive keratectomy (PRK), laser in situ keratomileusis (LASIK), and radial keratotomy (RK) with good success.
  Bandage contact lenses have also been used in studies in Europe through ophthalmology clinics to treat traumatic corneal abrasions with excellent results. A British study from 1987, found that large diameter contact lenses can be fitted satisfactorily without the use of special equipment such as keratometry. Studies in rabbits have also been performed showing improved rates of healing when using bandage contact lenses. BCLs have been used to treat epithelial defects from various causes for up to 7 months at a time.
  Arms: Group 2
Drug: Eyedrop — Fluoroquinolone eyedrops 4x/day
Drug: Hydrocodone — Hydrocone 1-2 tabs 4x/day if needed

SUMMARY:
Two percent of all patients presenting to the Emergency Departments have complaints involving the eye. Corneal abrasions are a common diagnosis with patients with eye pain and often cause significant discomfort. Current treatment includes a thorough evaluation of the eye followed by patching, empiric antibiotics, cycloplegics and oral pain medicines. This study will be a randomized controlled trial to determine the safety and efficacy of BCLs. It will involve the initial patient evaluation followed by a return visit to the Emergency Department within 36 hours for re-examination. At each visit, the patient will be assessed for the size and location of the abrasion along with their report of pain using a visual analog scale. Data will be recorded on a standard data collection sheet. Telephone contact will be made at 30 days to ensure resolution of abrasion and that no complications ensued.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ages 18-65 years who present to the emergency department.
* Traumatic corneal abrasion not associated with contact lens use or communicating or adjacent wounds to the eye.

Exclusion Criteria:

* Pregnant women
* Breast-feeding women
* Corneal abrasion associated with the wearing contact lenses
* Evidence of corneal ulcer, glaucoma or other ocular pathology, monocular vision
* Wound healing deficits such as collagen vascular disease or concomitant steroid use
* Use of other ocular medications, dry eyes, blepharitis
* Systemic infections
* Known allergies to medicines used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain scale | 24 hours post treatment
  The pain difference using Visual Analogue Scale

SECONDARY OUTCOMES:
Corneal defect size | 24 hours post treatment
  Reduction in size (mm) of the defect
Pain medication needed | 24 hours post treatment
  The amount of pain medication needed

CONTACTS AND LOCATIONS:
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.